CLINICAL TRIAL: NCT07219095
Title: Use of a Mental Health App in the Recovery of Adolescent Dancers From a Lower Extremity Injury: A Randomized Controlled Trial
Brief Title: Dance Mental Health App
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Sanford Scholars Program Mentor Funding (Unknown)
Responsible Party: Principal Investigator, Emily Cidambi, Orthopedic Surgeon, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 812643
Record Dates: First submitted 2025-08-25; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Ankle Injury; Foot Injury; Lower Extremity Injury
Keywords: dance; self-compassion
MeSH Terms: conditions — Ankle Injuries; Foot Injuries

STUDY DESIGN:
Intervention Model Description: Concurrent mental health intervention with the SuperBetter app synchronously with physical therapy rehab from a lower extremity injury in dancers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SuperBetter Arm (Experimental): Those randomized into the treatment group will be completing gamified mental health exercises in an app called SuperBetter for 10 minutes, 5 days per week, for 12 weeks alongside physical therapy.
  Interventions: Device: Mental Health App
- Control Arm (No Intervention): Those randomized into the observation group need only attend their physical therapy appointments and complete the questionnaires but will not use the mental health app.

INTERVENTIONS:
Device: Mental Health App — Participants will use the SuperBetter mobile app to participate in gamified mental health activities 5 days per week, 10 minutes per day, for 12 weeks alongside their physical therapy.
  Arms: SuperBetter Arm

SUMMARY:
This project aims to enhance self-compassion in adolescent dancers recovering from a foot and ankle injury by incorporating the use of a mental health intervention app using gamified design during their recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent (adult participant), or consent of parent/legal guardian in conjunction with adolescent assent (minor participant)
2. 13 to 18 years of age
3. Endorses dance as their primary sport, or participates 3 days per week or greater in dance prior to injury
4. Stated willingness to comply with all study procedures including the intervention regimen and availability for the duration of the study
5. Access to a device with which the SuperBetter app can be downloaded and used

Exclusion Criteria:

1. Dance is not a primary sport or less than 3 days per week spent dancing prior to injury (skater, gymnast, other sport)
2. Requiring surgery or prior surgery for the injury being treated
3. Injury outside of the leg below the knee
4. Known eating disorder or bone density issue (documented abnormal Z score and/or eating disorder diagnosis upon review of the medical chart)
5. Verbalized plans to not return to dance after recovery from the injury

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2029-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Number (or percentage) of participants who have returned to full, unrestricted dance after injury | 3, 6 and 12 months.
  Will be assessed as part of the clinical exam by asking current return to dance status

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Measures of Pediatric Anxiety, Depressive Symptoms, Pain Interference, and Mobility questionnaire | enrollment, 3 months, 6 months, 12 months, 18 months, and 24 months
  PROMIS scores for Emotional distress (anxiety and depression) and Pain interference subscales. Higher score and higher standard deviation from the norm are considered poorer function/worse outcomes.
Self Compassion Scale (SCS) - Short Form questionnaire | enrollment, 3 months, 6 months, 12 months, 18 months, and 24 months
  1 is the lowest possible overall calculated score, and the highest overall calculated score is 5, with greater scores indicating greater level of self-compassion.
Foot and Ankle Ability Measure (FAAM) Activities of Daily Living subscale and Sports Subscale questionnaire | enrollment, 3 months, 6 months, 12 months, 18 months, and 24 months
  Minimum calculated score for each subscale is 0% and highest score is 100% with the higher score meaning better function.

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Likely not relevant or needed by other centers at this time

REFERENCES:
- [Background] Christino MA, Fantry AJ, Vopat BG. Psychological Aspects of Recovery Following Anterior Cruciate Ligament Reconstruction. J Am Acad Orthop Surg. 2015 Aug;23(8):501-9. doi: 10.5435/JAAOS-D-14-00173. PMID 26209145
- [Background] Gennarelli SM, Brown SM, Mulcahey MK. Psychosocial interventions help facilitate recovery following musculoskeletal sports injuries: a systematic review. Phys Sportsmed. 2020 Nov;48(4):370-377. doi: 10.1080/00913847.2020.1744486. Epub 2020 Mar 25. PMID 32186423
- [Background] Walter HJ, Bukstein OG, Abright AR, Keable H, Ramtekkar U, Ripperger-Suhler J, Rockhill C. Clinical Practice Guideline for the Assessment and Treatment of Children and Adolescents With Anxiety Disorders. J Am Acad Child Adolesc Psychiatry. 2020 Oct;59(10):1107-1124. doi: 10.1016/j.jaac.2020.05.005. Epub 2020 May 18. PMID 32439401
- [Background] Neff KD, Toth-Kiraly I, Yarnell LM, Arimitsu K, Castilho P, Ghorbani N, Guo HX, Hirsch JK, Hupfeld J, Hutz CS, Kotsou I, Lee WK, Montero-Marin J, Sirois FM, de Souza LK, Svendsen JL, Wilkinson RB, Mantzios M. Examining the factor structure of the Self-Compassion Scale in 20 diverse samples: Support for use of a total score and six subscale scores. Psychol Assess. 2019 Jan;31(1):27-45. doi: 10.1037/pas0000629. Epub 2018 Aug 20. PMID 30124303
- [Background] Worthen-Chaudhari L, McGonigal J, Logan K, Bockbrader MA, Yeates KO, Mysiw WJ. Reducing concussion symptoms among teenage youth: Evaluation of a mobile health app. Brain Inj. 2017;31(10):1279-1286. doi: 10.1080/02699052.2017.1332388. Epub 2017 Jun 30. PMID 28665690
- [Background] Psihogios AM, Stiles-Shields C, Neary M. The Needle in the Haystack: Identifying Credible Mobile Health Apps for Pediatric Populations during a Pandemic and beyond. J Pediatr Psychol. 2020 Nov 1;45(10):1106-1113. doi: 10.1093/jpepsy/jsaa094. PMID 33068424
- [Background] Semenchuk BN, Strachan SM, Fortier M. Self-Compassion and the Self-Regulation of Exercise: Reactions to Recalled Exercise Setbacks. J Sport Exerc Psychol. 2018 Feb 1;40(1):31-39. doi: 10.1123/jsep.2017-0242. Epub 2018 Mar 26. PMID 29580155
- [Background] Neff KD, Bluth K, Toth-Kiraly I, Davidson O, Knox MC, Williamson Z, Costigan A. Development and Validation of the Self-Compassion Scale for Youth. J Pers Assess. 2021 Jan-Feb;103(1):92-105. doi: 10.1080/00223891.2020.1729774. Epub 2020 Mar 3. PMID 32125190
- [Background] Bantjes J, Hunt X, Cuijpers P, Kazdin AE, Kennedy CJ, Luedtke A, Malenica I, Petukhova M, Sampson N, Zainal NH, Davids C, Dunn-Coetzee M, Gerber R, Stein DJ, Kessler RC. Comparative effectiveness of remote digital gamified and group CBT skills training interventions for anxiety and depression among college students: Results of a three-arm randomised controlled trial. Behav Res Ther. 2024 Jul;178:104554. doi: 10.1016/j.brat.2024.104554. Epub 2024 May 3. PMID 38714104
- [Background] Noh YE, Morris T, Andersen MB. Psychological intervention programs for reduction of injury in ballet dancers. Res Sports Med. 2007 Jan-Mar;15(1):13-32. doi: 10.1080/15438620600987064. PMID 17365949
- [Background] van Winden D, van Rijn RM, Savelsbergh GJP, Oudejans RRD, Stubbe JH. The Association Between Stress and Injury: A Prospective Cohort Study Among 186 First-Year Contemporary Dance Students. Front Psychol. 2021 Nov 5;12:770494. doi: 10.3389/fpsyg.2021.770494. eCollection 2021. PMID 34803856

DOCUMENTS (1):
  • Study Protocol (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT07219095/Prot_000.pdf